CLINICAL TRIAL: NCT02072031
Title: A Randomized, Positive-controlled, Multicenter, Phase II Study of Anlotinib(AL3818) in Patients With Advanced Renal Cell Carcinoma(RCC)
Brief Title: Phase II Study of Anlotinib Versus Sunitinib in Patients With Advanced Renal Cell Carcinoma（RCC）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-06-IIA
Record Dates: First submitted 2014-01-20; First posted 2014-02-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Anlotinib; RCC
Keywords: Anlotinib; Sunitinib; Renal Cell Carcinoma（RCC）
MeSH Terms: interventions — anlotinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anlotinib (Experimental): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib
- Sunitinib maleate (Active Comparator): Sunitinib 50 mg qd p.o., 4 weeks out of 6.The treatment continued until disease progression or intolerable toxicity happened or patients withdrawal of consent.
  Interventions: Drug: Sunitinib maleate

INTERVENTIONS:
Drug: Anlotinib — Anlotinib p.o. qd
  Arms: Anlotinib
Drug: Sunitinib maleate — Sunitinib 50 mg p.o. qd
  Arms: Sunitinib maleate

SUMMARY:
Anlotibib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2、VEGFR3、PDGFRβ and c-Kit. It has the obvious resistance to new angiogenesis. The trial is to compare the efficacy and safety profile between Anlotinib and Sunitinib in patients with advanced Renal Cell Carcinoma(RCC).

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with histologically confirmed advanced renal cell carcinoma including clear cell component and not available for surgery
* 2.Without drug treatment for RCC or chemotherapy/cytokine therapy failure or resistant patients)
* 3.With measurable disease (using RECIST1.1)
* 4.18-75years,ECOG PS:0-1,Life expectancy of more than 3 months
* 5.Other cytotoxic drugs,radiation therapy,or surgery≥4 weeks
* 6.main organs function is normal
* 7.Signed and dated informed consent

Exclusion Criteria:

* 1.Previously received targeted therapy of the metastatic renal cell carcinoma (such as sunitinib, Sorafenib)
* 2.patients has many influence factors toward oral medications
* 3.Known brain metastases
* 4.patients with severe and failed to controlled diseases,including: suboptimal blood pressure control;suffering from myocardial ischemia or above grade I myocardial infarction, arrhythmias and Class I heart failure;activity or failure to control severe infections;liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis;poorly controlled diabetes (FBG)>10mmol/L);urine protein≥++,etc.
* 5.patients failed to heal wounds or fractures for Long-term
* 6.patients occurred venous thromboembolic events within 6 months
* 7.patients has HIV-positive or organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | each 42 days up to PD or death(up to 36 months)
  The PFS time is defined as time from randomization to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of: "death", "last tumor assessment", "last follow up date" or "last date in drug log".

SECONDARY OUTCOMES:
Objective Response Rate | each 42 days up to intolerance the toxicity or PD (up to 36 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule by enhanced CT/MRI scan every two cycles or Sunitinib maleate by enhanced CT/MRI scan every cycle. Objective Response Rate (ORR) is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 36 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule by enhanced CT/MRI scan every two cycles or Sunitinib maleate by enhanced CT/MRI scan every cycle. Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).
Overall Survival (OS) | From randomization until death (up to 36 months)
  OS was defined as time from date of randomization to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi medical university affiliated tumor hospital, Nanning, Guangxi
  - Harbin medical university affiliated tumor hospital, Haerbin, Heilongjiang
  - The 81st Hospital of Chinese PLA, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - China General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Liaoning Province Tumor Hospital, Shenyang, Liaoning
  - Qilu Hospital，Shandong University, Jinan, Shandong
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Lin J, Fang Q, Zheng X. Cost-effectiveness analysis of anlotinib versus sunitinib as first-line treatment for metastatic renal cell carcinoma in China. PLoS One. 2023 Feb 7;18(2):e0281402. doi: 10.1371/journal.pone.0281402. eCollection 2023. PMID 36749752
- See also: NLM — http://www.nlm.nih.gov/medlineplus/
- See also: Druginfo — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: Sunitinib — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0341031547&QV1=SUNITINIB+MALATE